CLINICAL TRIAL: NCT01689974
Title: Phase II Randomized Trial of Ipilimumab Versus Ipilimumab and Radiotherapy in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated because PI left institution. Planned Statistical analysis not available
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-02746
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; Radiation Therapy; Immunology; Abscopal
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Ipilimumab (Other): Ipilimumab administered alone Day 4, 25, 46, and 67
  Interventions: Drug: Ipilimumab
- Arm B: Ipilimumab and Radiation (Other): Radiation Therapy and Ipilimumab. Radiation treatment is administered for 5 fractions (sessions) over 1 week. On Day 4 treatment with Ipilimumab begins and continues on Days 25, 46, and 67.
  Interventions: Drug: Ipilimumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab will be administered alone on day 4, 25, 46 and 67.
  Other Names: Yervoy
Radiation: Radiation Therapy — Radiation is given over one week interval On the fourth day of radiation (day 4)Ipilimumab is administered and repeated on Days 25, 46 and 67.
  Arms: Arm B: Ipilimumab and Radiation

SUMMARY:
An attractive area of research regards immune manipulations to recover some of the patient's immune response to his/her tumor, a strategy that has the advantages of being both natural and potentially long-lasting.[1] We propose to combine immunotherapy with radiotherapy directed to a metastatic site, to create a "hub" for in vivo immunization to the tumor, to enable "tumor rejection" at the other metastatic sites. This "in vivo immunization" is explored as a viable alternative to an individualized vaccine approach. Preclinical data generated by us and others support a "proof of principle" clinical trial that may open the field to an alternative use of radiotherapy in a novel partnership with cancer immunotherapy.[2]

DETAILED DESCRIPTION:
In addition, we propose to perform immune-monitoring of the patients accrued to the trial to generate important information for hypothesis-driven research about the mechanisms behind the clinical findings, to be tested in the laboratory.

An attractive area of research regards immune manipulations to recover some of the patient's immune response to his/her tumor, a strategy that has the advantages of being both natural and potentially long-lasting.[1] We propose to combine immunotherapy with radiotherapy directed to a metastatic site, to create a "hub" for in vivo immunization to the tumor, to enable "tumor rejection" at the other metastatic sites. This "in vivo immunization" is explored as a viable alternative to an individualized vaccine approach. Preclinical data generated by us and others support a "proof of principle" clinical trial that may open the field to an alternative use of radiotherapy in a novel partnership with cancer immunotherapy.[2]

In addition, we propose to perform immune-monitoring of the patients accrued to the trial to generate important information for hypothesis-driven research about the mechanisms behind the clinical findings, to be tested in the laboratory.

The specific aims of the study are:

1. To explore the induction of immunity-mediated tumor response outside the radiation field (abscopal effect) after radiation/Ipilimumab in metastatic melanoma, by estimating and comparing response rates in patients treated with Ipilimumab alone (Arm A) versus ipilimumab and radiation (Arm B).
2. To compare the induction of a T-cell response in patients with metastatic melanoma treated with either ipilimumab alone or in combination with radiation.

All patients with metastatic melanoma with at least 2 measurable sites of disease are eligible. Extent of metastatic disease is recorded by CT scanning or MRI before therapy. Patients will then be randomized to Ipilimumab 3 mg/kg IV over 90 minutes alone versus Ipilimumab 3 mg/kg IV over 90 minutes plus radiotherapy to one of their measurable lesions, 6 Gy delivered daily x 5 days (Monday through Friday) (conformally or by IMRT/IGRT, to maximally spare normal tissue), for a total of 30 Gy. For patients assigned to the Ipilimumab/RT arm, Ipilimumab treatment starts after radiotherapy, with a dose given on day 4 from the first radiotherapy fraction. All patients will then have ipilimumab infusions repeated on Days 25, 46 and 67. Patients will be re-imaged (CT imaging or MRI) on Week 12 and evaluated for response (defined as an objective response of another metastatic site outside the radiation field).

The main immunological end-point will be the induction or boosting of treatment induced T cells (CD4+ and CD8+) and B cells for defined antigen approaches. In addition, the magnitude and duration of T- and B-cell responses will be examined. Treatment-induced responses will be calculated as the difference between the pre-treatment measurement and the measurement at the different time points at which blood will be collected (time of evaluation) in the same patient. The percentage of patients with the induction of treatment-induced T- and B-cell responses will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document;
* Histologic diagnosis of locally unresectable, metastatic melanoma.
* Any BRAF status is permitted
* Any prior therapy is permitted except prior therapy with ipilimumab.
* Patients must have at least 2 distinct measurable metastatic sites, with one of at least 1 cm or larger in its largest diameter and may have additional non-measurable but established metastatic lesions (i.e. bone metastases).
* Patients must have adequate organ and marrow function as defined by initial laboratory tests:

  * WBC 2000/uL
  * ANC 1000/uL
  * Platelets 50 x 103/uL
  * Hemoglobin 8 g/dL
  * Creatinine 3.0 x ULN
  * AST/ALT 2.5 x ULN for patients without liver metastasis
  * Bilirubin 3.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL;
* Performance status ECOG 0-1 or Karnofsky > 50%;
* Men and women, ages > 18 year old of age;
* Life expectancy > 3 months
* Stable brain metastases for at least 4 weeks and not steroid dependent;
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study.

Exclusion Criteria:

* Patients having no lesions outside the field of radiation thus nullifying the ability to measure an abscopal effect;
* Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis;
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea;
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab);
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids;
* Women who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 8 weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding;
* Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after study drug is stopped;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia C. Formenti, M.D., Principal Investigator — NYULMC Department Radiation Oncology
Locations (1):
- NYU Clinical Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Ipilimumab and Radiation: Radiation Therapy and Ipilimumab. Radiation treatment is administered for 5 fractions (sessions) over 1 week. On Day 4 treatment with Ipilimumab begins and continues on Days 25, 46, and 67.
  Radiation Therapy and Ipilimumab: Radiation is given over one week interval On the fourth day of radiation (day 4)Ipilimumab is administered and repeated on Days 25, 46 and 67.
Period: Overall Study
Arm/Group | Arm A: Ipilimumab | Arm B: Ipilimumab and Radiation
Started | 5 | 5
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — Termination of Study | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ipilimumab | Arm B: Ipilimumab and Radiation | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Response Rates of Ipilimumab Alone and of Ipilimumab With Radiation Therapy and to Estimate the Difference Between Response Rates With Ipilimumab Alone and Ipilimumab With Radiation Therapy
Description: Eligible patients have metastatic melanoma with at least 2 measurable sites of disease. All patients with metastatic melanoma are eligible to be randomly assigned to Ipilimumab 3mg/kg IV over 90 minutes versus Ipilimumab 3 mg/kg IV over 90 minutes and radiotherapy to one of their measurable lesions, 6 Gy X5 (conformally or by IMRT/IGRT, to maximally spare normal tissue). For patients assigned to the Ipi/RT arm, Ipilimumab treatment starts after radiotherapy, with a dose given on day 4 from the first radiotherapy fraction and repeated on Days 25, 46 and 67. Patients will be re-imaged on Week 12 and evaluated for response (defined as an objective response of another metastatic site outside the radiation field). This response will be evaluated assessing clinical and CT responses in the non-irradiated measurable metastatic sites.
Time Frame: 2 years
Population: Study terminated because PI left institution. Data cannot be reported because 2 year data were not collected and were not analyzed.
Arm/Group | Arm A: Ipilimumab | Arm B: Ipilimumab and Radiation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A: Ipilimumab | Arm B: Ipilimumab and Radiation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes